CLINICAL TRIAL: NCT05607004
Title: A Phase 2 Trial of (Z)-Endoxifen + Goserelin as Neoadjuvant Treatment for Premenopausal Women With ER+, HER2-, Breast Cancer
Brief Title: (Z)-Endoxifen for the Treatment of Premenopausal Women With ER+/HER2- Breast Cancer
Acronym: EVANGELINE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Atossa Therapeutics, Inc. (Industry)
Collaborators: InClin (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATOS-Z-201
Record Dates: First submitted 2022-10-26; First posted 2022-11-07 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Breast Neoplasms; Invasive Breast Cancer; Estrogen-receptor-positive Breast Cancer; HER2-negative Breast Cancer
Keywords: breast cancer; ER+/HER2-; endocrine therapy; neoadjuvant; (Z)-endoxifen; exemestane; goserelin; Ki-67; estrogen receptor negative; human epidermal growth factor receptor 2 negative; Stage II; tamoxifen; PKCB1
MeSH Terms: conditions — Breast Neoplasms | interventions — 4-hydroxy-N-desmethyltamoxifen; Goserelin

STUDY DESIGN:
Intervention Model Description: This multicenter open-label study consists of two cohorts: PK and Treatment
  The PK Cohort is a dose finding study to identify the dose to use in the Treatment Cohort.
  The Treatment Cohort includes a single treatment arm. All participants will be assigned to (Z)-endoxifen + goserelin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PK Cohort (Experimental): (Z)-endoxifen capsules orally once daily for 4 weeks. Initial (Z)-endoxifen dose evaluated will be 40 mg with an option to evaluate 20 mg or 80 mg.
  The PK Cohort participants may extend treatment based on Ki-67% at Week 4.
  If Ki-67 ≤ 10% at Week 4, participant will be offered option to continue on this treatment for up to 6 cycles/Week 24. Each cycle is 28 days.
  If Ki-67 > 10% at Week 4, participant will be withdrawn and go on to surgery.
  Interventions: Drug: (Z)-endoxifen
- Treatment Cohort - Single Treatment Arm (Experimental): (Z)-endoxifen 40mg capsules orally once daily for 4 weeks + goserelin 3.6 mg by subcutaneous implant approximately every 28 days. (Z)-endoxifen 40mg dose based on results of PK Cohort.
  If Ki-67 ≤ 10% at Week 4, continue on this treatment for up to 6 cycles/Week 24. Each cycle is 28 days. And then go on to surgery within 3 weeks of Cycle 6 day 26.
  If Ki-67 > 10% at Week 4, participant will complete early termination assessments.
  Interventions: Drug: (Z)-endoxifen; Drug: goserelin
- PK Cohort 80 mg (Experimental): (Z)-endoxifen 80 mg capsules orally once daily for 4 weeks.
  The PK Cohort participants may extend treatment based on Ki-67% at Week 4.
  If Ki-67 ≤ 10% at Week 4, participant will be offered option to continue on this treatment for up to 6 cycles/Week 24. Each cycle is 28 days.
  If Ki-67 > 10% at Week 4, participant will be withdrawn and go on to surgery.
  Interventions: Drug: (Z)-endoxifen
- PK Cohort 80 mg + OFS (Experimental): (Z)-endoxifen 80 mg capsules orally once daily for 4 weeks + goserelin 3.6 mg by subcutaneous implant approximately every 28 days.
  The PK Cohort participants may extend treatment based on Ki-67% at Week 4.
  If Ki-67 ≤ 10% at Week 4, participant will be offered option to continue on this treatment for up to 6 cycles/Week 24. Each cycle is 28 days.
  If Ki-67 > 10% at Week 4, participant will be withdrawn and go on to surgery.
  Interventions: Drug: (Z)-endoxifen; Drug: goserelin

INTERVENTIONS:
Drug: (Z)-endoxifen — (Z)-endoxifen capsules. Doses of (Z)-endoxifen to be evaluated include 20 mg (two x 10 mg capsules), 40 mg (one 40 mg capsule) and 80 mg (two x 40 mg capsules).
  Other Names: endoxifen
Drug: goserelin — goserelin 3.6 mg subcutaneous implant
  Other Names: Zoladex
  Arms: PK Cohort 80 mg + OFS; Treatment Cohort - Single Treatment Arm

SUMMARY:
This open-label research study is studying (Z)-endoxifen as a possible treatment for pre-menopausal women with ER+/HER2- breast cancer. (Z)-endoxifen belongs to a group of drugs called selective estrogen receptor modulators or "SERM", which help block estrogen from attaching to cancer cells. This study has two parts: a pharmacokinetic part and a treatment part.

The PK part (how the body processes the drug) will enroll about 18 participants. All participants will take (Z)-endoxifen capsules daily. Twelve participants will be randomly assigned (50/50 chance) to take (Z)-endoxifen alone or (Z)-endoxifen with a monthly injection of goserelin a drug that temporarily stops the ovaries from making estrogen. This part will help determine the best dose of (Z)-endoxifen by measuring the drug levels in the blood and how long the body takes to remove it.

The Treatment Cohort has been simplified to a single study arm (Z)-endoxifen + goserelin. Up to 20 participants will be enrolled that have a baseline Ki-67 ≤ 10% and 45 participants will be enrolled that have a baseline Ki-67>10%.

A key goal of the study is to see if (Z)-endoxifen can slow down or stop tumor growth as measured by a reduction in Ki-67 levels. Tumor tissue samples will be taken by breast biopsy after about 4 weeks of treatment to check levels of this biomarker. If the tumor shows signs of response, participants can continue treatment for up to 24 weeks or until they have surgery.

Study participation is up to 6 months (24 weeks of treatment) followed by surgery and a one-month follow up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Female sex assigned at birth. Female to male transgender individuals who have not had any hormonal therapy may be considered for the trial after review and approval from the medical monitor and study sponsor.
2. Age 18 years or older
3. Not lactating, pregnant, or planning to become pregnant in the next year and agrees to take adequate steps to prevent becoming pregnant beginning at informed consent, during treatment and for 9 months after last dose and agree to not breast feed during treatment and for 3 months after last dose.
4. Must agree to use at least one non-hormonal highly effective method of contraception for the entire duration of study participation beginning at informed consent. Highly effective methods of birth control are defined as those, alone or in combination, that resulted in a low failure rate of <1% per year when used consistently and correctly such as intrauterine devices (IUDs, non-hormonal such as copper IUD), bilateral tubal occlusion, sexual abstinence or vasectomized partner
5. Premenopausal defined as any female who:

   1. is menstruating or
   2. is not menstruating (last menstrual period > 3 months prior to registration) but has a plasma estradiol in the premenopausal range as assessed locally
6. Pathologic confirmation of strongly estrogen receptor positive (ER+) (defined as estrogen receptor [ER] ≥ 67% or Allred Score 6-8) by local institution protocol
7. Eastern Cooperative Oncology Group ECOG Performance Status (ECOG PS) of 0 to 2
8. Nottingham (Elston-Ellis) Grade 1 or 2
9. HER2- breast cancer (histologically confirmed) using American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines
10. Clinical T2 or T3 invasive breast cancer (per American Joint Committee on Cancer [AJCC] 8th edition clinical staging)
11. Clinical N0 or N1 invasive breast cancer (per American Joint Committee on Cancer [AJCC] 8th edition clinical staging)
12. MRI ≤ 35 days of registration
13. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects
14. Willing to provide blood and breast tissue samples for research purposes at specified timepoints for the duration of their participation in the trial.

Exclusion Criteria:

1. Bilateral invasive breast cancer; Inflammatory breast cancer defined as clinically significant erythema of the breast and/or documented dermal lymphatic invasion or bilateral invasive breast cancer (patients with pre-malignant disease or DCIS/LCIS in contralateral breast are eligible)
2. Prior diagnosis or treatment for breast cancer, including carcinoma in situ, or history of any other active malignancy within the past 2 years prior to study entry with the exception of:

   1. Adequately treated in situ carcinoma of the cervix uteri
   2. Adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin
   3. Any other malignancy with a life expectancy of less than 2 years
3. Any uncontrolled intercurrent illness including, but not limited to:

   1. Ongoing or active infection requiring systemic treatment with strong inhibitors/inducers of CYP450 enzymes (including bacterial infection, fungal infection, or detectable viral infection).
   2. Symptomatic congestive heart failure,
   3. Unstable angina pectoris,
   4. Uncontrolled symptomatic cardiac arrhythmias
   5. Uncontrolled hypertension
   6. Uncontrolled diabetes (Hemoglobin A1c [HbA1c] >7%)
   7. Marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval > 470 milliseconds [msec]) using Fridericia's QT correction formula seen ≤ 28 days of registration
4. Any of the following co-morbid conditions:

   1. Known cataracts or retinopathy
   2. History of deep vein thrombosis (DVT)/pulmonary embolism (PE)
   3. Known activated protein C (APC) resistance, an inherited coagulation disorder
   4. End stage kidney disease requiring dialysis
5. Evidence of the following laboratory abnormalities ≤ 28 days prior to registration:

   1. Total bilirubin ≥ 1.5 x upper limit of normal (ULN)
   2. Aspartate aminotransferase (AST) or alanine amino transferase (ALT) ≥ 2.5 x ULN
   3. Platelet count (PLT) ≤ 75,000/mm3
   4. Hemoglobin (Hb) ≤ 10 g/dL
6. Hormonal therapies including birth control and hormone replacement therapy, or prior use of androgen-based therapy during the study or within 1 week of registration. If subject has a prior medical history of Depo-Provera®, it is recommended that the last dose of 3-month contraceptive agents are > 2.5 months from registration.
7. Allergy to endoxifen, goserelin, or exemestane or any of their components
8. Participation in another investigational clinical trial ≤ 6 months of registration
9. Known metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female sex assigned at birth
Enrollment: 87 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
PK Cohort - (Z)-endoxifen steady-state plasma concentrations | After 4 weeks of treatment
  (Z)-endoxifen steady-state plasma concentrations (Css) of evaluable subjects who completed at least one cycle of treatment (28 +/- 3 days)
For Analysis of Cohort A (Treatment Cohort): determine whether the week 4 Ki-67≤10% rate is at least 65% | After 4 weeks of treatment
  For analysis Cohort A (subjects that have a baseline Ki-67>10%): the primary objective is to determine whether the Week 4 Ki-67 ≤ 10% rate is at least 65% among premenopausal women with primary estrogen receptor positive (ER+), Human Epidermal Growth Factor Receptor 2 negative (HER2-) breast cancer.
For analysis Cohort B (Treatment Cohort): determine the objective tumor response rate at 24 weeks | After 24 weeks of treatment
  For analysis Cohort B (subjects have baseline Ki-67≤ 10%): the primary objective is to determine the objective tumor response rate at 24 weeks among premenopausal women with ER+, HER2-, Ki-67 ≤ 10% breast cancer receiving (Z) endoxifen plus goserelin.

SECONDARY OUTCOMES:
PK Cohort - Area under the plasma (Z)-endoxifen concentration-time curve from time zero to last measurable concentration | Days 1 and 28
  Area under the plasma (Z)-endoxifen concentration-time curve from time zero to last measurable concentration (AUC0-24) on Days 1 and 28 of evaluable subjects who completed at least one cycle of treatment (28 +/- 3 days)
PK Cohort - Area under the plasma (E)-endoxifen concentration-time curve from time zero to last measurable concentration | Days 1 and 28
  Area under the plasma (E)-endoxifen concentration-time curve from time zero to last measurable concentration (AUC0-24) on Days 1 and 28 of evaluable subjects who completed at least one cycle of treatment (28 +/- 3 days)
PK Cohort - Accumulation and accumulation half-life | Days 1 and 28
  Accumulation and accumulation half-life (Day 28 AUC0-24/Day 1 AUC0-24) of evaluable subjects who completed at least one cycle of treatment (28 +/- 3 days)
PK Cohort - (Z)-endoxifen steady-state clearance | up to 28 days
  (Z)-endoxifen CLss (steady-state clearance) of evaluable subjects who completed at least one cycle of treatment (28 +/- 3 days)
PK Cohort - (E)-endoxifen steady-state clearance | up to 28 days
  (E)-endoxifen CLss (steady-state clearance) of evaluable subjects who completed at least one cycle of treatment (28 +/- 3 days)
PK Cohort - Maximum plasma (Z)-endoxifen concentration | up to 28 days
  Maximum plasma (Z)-endoxifen concentration (Cmax) of evaluable subjects who completed at least one cycle of treatment (28 +/- 3 days)
PK Cohort - Maximum plasma (E)-endoxifen concentration | up to 28 days
  Maximum plasma (E)-endoxifen concentration (Cmax) of evaluable subjects who completed at least one cycle of treatment (28 +/- 3 days)
PK Cohort - Time to plasma (Z)-endoxifen maximum concentration | up to 28 days
  Time to plasma (Z)-endoxifen maximum concentration (Tmax) of evaluable subjects who completed at least one cycle of treatment (28 +/- 3 days)
PK Cohort - Time to plasma (E)-endoxifen maximum concentration | up to 28 days
  Time to plasma (E)-endoxifen maximum concentration (Tmax) of evaluable subjects who completed at least one cycle of treatment (28 +/- 3 days)
PK Cohort - plasma (Z)-endoxifen concentration | Day 1 up to 12 weeks and up to end of treatment or up to 24 weeks.
  Trough concentrations of (Z)-endoxifen for subjects in the Treatment Extension
PK Cohort - plasma (E)-endoxifen concentration | Day 1 up to 12 weeks and up to end of treatment or up to 24 weeks.
  Trough concentrations of (Z)-endoxifen for subjects in the Treatment Extension
PK Cohort- Endocrine sensitive disease rate based on Ki-67 percent after 4 weeks of treatment | After 4 weeks of treatment
  Endocrine sensitive disease rate will be estimated as the percentage of subjects whose 4-week tumor biopsy finds Ki-67 less than or equal to 10 percent among evaluable subjects who began protocol treatment
All Cohorts - Incidence and severity of adverse events per CTCAE by treatment | Informed consent up to follow up visit or up to 30 weeks
  Incidence and severity of adverse events per CTCAE
All Cohorts - Incidence of Serious Adverse Events assessed by CTCAE version 5.0 | Informed consent up to follow up visit or up to 30 weeks
  Serious adverse events and adverse events leading to discontinuation of neoadjuvant treatment
All Cohorts - Incidence of Dose Reductions | Informed consent up to end of treatment or up to 24 weeks
  The incidence of dose reductions
All Cohorts - Change in estradiol and estrone | Day 1, up to 4 weeks and up to end of treatment or up to 24 weeks.
  Percent change from baseline in E1 and E2 at 4 weeks, and 24 weeks
All Cohorts - Percentage of subjects whose serum thymidine kinase 1 (TK1) is not detectable at 4 weeks and 24 weeks. | Day 1, up to 4 weeks and up to end of treatment or up to 24 weeks.
  Percent of subjects whose serum TK1 is not detectable at 4 weeks and 24 weeks
Treatment Cohorts - Assess additional PK parameters of (Z)-endoxifen and (E)-endoxifen | Day 1, up to 4 weeks, up to 12 weeks and up to 24 weeks
  Tissue and plasma (Z)-endoxifen and (E)-endoxifen concentrations at 4 weeks and 24 weeks
Treatment Cohorts - Radiographic Response Rate in the breast | Baseline Assessment, up to 4 weeks, up to 12 weeks, and up to 24 weeks
  Radiographic response rate in the breast at 4, 12, and 24 weeks as assessed by RECIST 1.1 criteria
Treatment Cohorts - Pathologic Complete Response per American Joint Committee on Cancer staging system at time of surgery | At time of surgery or up to 27 weeks
  Pathologic Complete Response (pCR) at surgery defined as the absence of residual invasive breast cancer on hematoxylin and eosin evaluation of the resected breast specimen and of all sampled lymph nodes (sentinel ± axillary) removed following completion of neoadjuvant systemic therapy
Treatment Cohorts - Pre-Operative Endocrine Prognostic Index at time of surgery | At time of surgery or up to 27 weeks
  Rate of Pre-Operative Endocrine Prognostic Index (PEPI) 0 at time of surgery using residual tumor specimen
Treatment Cohorts - Residual Cancer Burden at time of surgery | At time of surgery or up to 27 weeks
  Rate of residual cancer burden class of 0-I at time of surgery
Treatment Cohorts - Conversion Rate | From baseline to time of surgery or up to 27 weeks
  Evaluate the conversion rate from breast conservation surgery ineligible to breast conservation surgery eligible. Evaluation is based on surgeon's impression of the type of surgery participant is eligible for (candidate for lumpectomy, candidate for modified radical mastectomy, inoperable) at baseline compared to surgeon's impression after completion of neoadjuvant treatment
Treatment Cohorts - Actual Conversion Rate | At time of surgery or up to 27 weeks
  Evaluate the actual rate of breast conservation surgery. Evaluation will be based on the extent of the surgical procedure at the time of surgery (lumpectomy, partial or segmental mastectomy, simple/total mastectomy, skin and/or nipple sparing mastectomy, radical mastectomy or other)
Treatment Cohorts - Change in menopause quality of life (MENQOL) | baseline, up to 4 weeks, and up to 24 weeks
  Evaluate changes in menopause symptoms after neoadjuvant treatment
Treatment Cohorts - Nodal response rate | At time of surgery or up to 27 weeks
  Rate of nodal pCR in subjects with biopsy proven nodal disease

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Goetz, MD, Principal Investigator — Mayo Clinic
Locations (15):
- United States (15):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - California Research Institute, Los Angeles, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Baylor University, Houston, Texas
  - Tranquility Research, Webster, Texas
  - Bon Secours Cancer Institute, Midlothian, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No